CLINICAL TRIAL: NCT03489018
Title: The Effect of Fractional Doses of Pneumococcal Conjugate Vaccines (PCV10 and PCV13) on Immunogenicity and Vaccine-serotype Carriage in Kenyan Infants
Brief Title: The Effect of Fractional Doses of Pneumococcal Conjugate Vaccines on Immunogenicity and Carriage in Kenyan Infants
Acronym: FPCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College, London (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); Bill and Melinda Gates Foundation (Other); National Institute of Health Research (NIHR) Mucosal Pathogens Research Unit (MPRU) (Unknown); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QA1075
Record Dates: First submitted 2018-03-29; First posted 2018-11-21 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2023-03

CONDITIONS: Pneumococcal Infection; Streptococcus Pneumoniae Infection; Invasive Pneumococcal Disease, Protection Against
Keywords: Pneumococcal Vaccines;; Immunogenicity, Vaccine; 10-valent pneumococcal vaccine; 13-valent pneumococcal vaccine; Schedule; Pneumococcal Infection; Kenya; Infant; Vaccines, Conjugate; Humans; Immunization schedule; Streptococcus pneumoniae; vaccine; Dose-Response Relationship, immunologic; Equivalence Trial as Topic
MeSH Terms: conditions — Pneumococcal Infections | interventions — 10-valent pneumococcal conjugate vaccine; PHiD-CV vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of seven groups for the duration of the study:
  A. Full dose PCV13 vaccination in a 2p+1 schedule; B. 40% fractional dose PCV13 vaccination in a 2p+1 schedule; C. 20% fractional dose PCV13 vaccination in a 2p+1 schedule; D. Full dose PCV10 vaccination in a 2p+1 schedule; E. 40% fractional dose PCV10 vaccination in a 2p+1 schedule; F. 20% fractional dose PCV10 vaccination in a 2p+1 schedule; G. Full dose PCV10 vaccination in a 3p+0 schedule.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, parents of participants and all of the study team apart from the vaccinator will be masked with respect to the infant's allocation to a trial arm between A-F. If randomly allocated to trial arm G, parents and study personnel will be unmasked due to the necessity for trial arm G to receive a different vaccine schedule compared to trial arms A-F. It is thought that this unmasking will have minimal impact on retention, follow up and outcome assessment across the trial arms for primary and secondary outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Full dose PCV13 (2p+1 schedule) (Active Comparator): Full dose PCV13 administration in 2p+1 schedule
  Interventions: Biological: PCV13
- 40% dose PCV13 (2p+1 schedule) (Experimental): Fractional (40%) dose PCV13 administration in 2p+1 schedule
  Interventions: Biological: PCV13
- 20% dose PCV13 (2p+1 schedule) (Experimental): Fractional (20%) dose PCV13 administration in 2p+1 schedule
  Interventions: Biological: PCV13
- Full dose PCV10 (2p+1 schedule) (Active Comparator): Full dose PCV10 administration in 2p+1 schedule
  Interventions: Biological: PCV10
- 40% dose PCV10 (2p+1 schedule) (Experimental): Fractional (40%) dose PCV10 administration in 2p+1 schedule
  Interventions: Biological: PCV10
- 20% dose PCV10 (2p+1 schedule) (Experimental): Fractional (20%) dose PCV10 administration in 2p+1 schedule
  Interventions: Biological: PCV10
- Full dose PCV10 (3p+0 schedule) (Active Comparator): The current vaccine (PCV10) and schedule (3p+0) in use in the Kenyan routine immunisation programme as an additional comparison arm.
  Interventions: Biological: PCV10

INTERVENTIONS:
Biological: PCV10 — Experimental arms will receive a lower dose of the intervention than the marketed dose.
  Other Names: Synflorix (GlaxoSmithKline plc.); 10-valent pneumococcal conjugate vaccine
  Arms: 20% dose PCV10 (2p+1 schedule); 40% dose PCV10 (2p+1 schedule); Full dose PCV10 (2p+1 schedule); Full dose PCV10 (3p+0 schedule)
Biological: PCV13 — Experimental arms will receive a lower dose of the intervention than the marketed dose.
  Other Names: Prevnar 13 (Pfizer Inc.); 13-valent pneumococcal conjugate vaccine; Prevnar13
  Arms: 20% dose PCV13 (2p+1 schedule); 40% dose PCV13 (2p+1 schedule); Full dose PCV13 (2p+1 schedule)

SUMMARY:
Before the introduction of pneumonia vaccines in 2000, between 700,000 - 1 million children died each year as a result of infection with the bacteria Streptococcus pneumoniae and the resulting diseases, namely, meningitis, sepsis and pneumonia. Most of the deaths were in Africa and Asia. Where the vaccines have been introduced, they have been highly effective and have already reduced disease. However, at 10 USD per child, they are not affordable to most low-income countries without financial support from Gavi, the Vaccine Alliance.

This project aims to assess whether lower doses of the two commercially available pneumonia vaccines can protect Kenyan infants as well as the full dose. The results could be used to increase the affordability of the pneumonia vaccine, and enable delivery of the vaccine to continue in the absence of Gavi support.

DETAILED DESCRIPTION:
Background:

PCV is currently the most expensive vaccine in the routine immunisation schedule in Gavi-supported countries. This study aims to provide evidence which may enable a substantial decrease in the cost of PCV programmes, therefore increasing the sustainability of PCV programmes in low and middle income countries (LMICs). We propose to assess whether fractional (20% and 40%) doses of pneumococcal conjugate vaccine (PCV10 and PCV13) in a 2p+1 schedule (2 primary doses followed by a booster dose) induce non-inferior immunogenicity and effects on vaccine-serotype carriage when compared to the full dose. These lower doses could convert new 4-dose vials of PCVs into 10- or 20-dose vials, ready for immediate implementation in LMIC programmes.

Primary objective:

Non-inferior immunogenicity at 1-month post-boost (10 months of age). Non-inferiority will be reached if the lower CI around the ratio of geometric mean concentrations (GMC) of IgG (fractional/full dose) is >0.5 (i.e. the 2-fold criterion).

Secondary objectives:

Non-inferior immunogenicity at 1-month post-primary series (18 weeks of age). Non-inferiority will be achieved if the lower limit of the 95% confidence interval (CI) around the difference in the proportion of 'responders', children with IgG>=0.35 mcg/ml, (fractional dose group - full dose group) is >-10% for at least 8 of the 10 vaccine types in the PCV10 arms and at least 10 of the 13 vaccine types in the PCV13 arms.

The opsonophagocytic activity of the antibody response to 7 serotypes after full/ fractional doses at the 1-month post-boost time point.

The direct vaccine effectiveness of full/fractional doses of PCV13 against carriage of serotypes 6A and 19A, with primary analyses at 18 months of age and secondary analyses at 9 months of age.

The proportion of children with evidence of vaccine-serotype carriage by trial arm at 9 and 18 months of age.

The geometric mean concentration (GMC) of serotype-specific IgG after the primary series of the 2p+1 schedule, prior to boost, at 9 months of age.

The geometric mean concentration (GMC) of serotype-specific IgG after three doses of vaccine in a 2p+1 schedule at 18 months of age.

The carriage prevalence at 9 and 18 months of age and IgG concentrations at 4 weeks after the primary series after full dose of PCV10 in a 3p+0 schedule, and full/ fractional doses of PCV10/13 in a 2p+1 schedule.

Trial design:

A phase IV individually-randomised controlled trial of full or fractional (20% or 40%) doses of PCV10/ PCV13, given as a 3-dose schedule to infants: 2 doses at 6 and 14 weeks of age and a booster dose at 9 months (the 2p+1 schedule) or 3 full doses at 6, 10 and 14 weeks of age (the 3p+0 schedule).

At 6-8 weeks of age, 300 infants will be enrolled at random into each of the seven trial arms and followed until 18 months of age.

The seven trial arms:

A. Full dose PCV13 vaccination in a 2p+1 schedule. B. 40% fractional dose PCV13 vaccination in a 2p+1 schedule. C. 20% fractional dose PCV13 vaccination in a 2p+1 schedule. D. Full dose PCV10 vaccination in a 2p+1 schedule. E. 40% fractional dose PCV10 vaccination in a 2p+1 schedule. F. 20% fractional dose PCV10 vaccination in a 2p+1 schedule. G. Full dose PCV10 vaccination in a 3p+0 schedule. This arm would represent the current vaccine and schedule in the Kenyan routine immunisation programme and would act as an additional comparison arm.

Study procedures:

No study procedures will be conducted without prior parental informed consent. Participants in trial arms A-F will provide 3 or 5 blood samples in the course of the trial at enrolment, 4 weeks post-primary series (approximately 18 weeks of age) and 4 weeks post-boost (approximately 10 months of age); additionally a random selection of half the participants will contribute blood samples pre-boost (9 months of age) and at the last study visit (18 months of age).

Participants in trial arm G will provide 2 blood samples (at enrolment and at 4 weeks post-primary series (approximately 18 weeks of age).

All participants will provide 2 nasopharyngeal swabs at approximately 9 and 18 months of age and contribute safety data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 6-8 weeks of age (HIV positive or negative but with no symptoms of current clinical immunosuppression i.e. HIV infection at WHO clinical stage 1);
* Parents are willing to provide informed consent for their child to participate in the study
* Parents and infant are likely to remain in the study area until the infant is 18 months of age and comply with study requirements including the requirement to return to the same health facility to obtain all other childhood vaccines.

Exclusion Criteria:

* Infants >8 weeks of age at time of enrolment
* Signs or symptoms of immunosuppression or HIV infection clinical stage 2 or above.
* Acute illness (e.g. febrile disease) on the day of vaccination
* Contraindications precluding vaccination (e.g. hypersensitivity to any component of the vaccine, including diphtheria toxoid)
* Previous PCV vaccination
* Family are planning to migrate out of the study areas before the end of the study follow-up
* Family are planning to obtain the subsequent vaccine doses of the routine immunisation schedule elsewhere and therefore their child may receive a full dose under the routine vaccination programme.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2100 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: The ratio of IgG GMCs at 1-month post boost | 4-weeks post-boost (approximately 10 months of age)
  The ratio of the geometric mean concentrations of IgG after vaccination with 3 full or fractional doses of PCV

SECONDARY OUTCOMES:
Immunogenicity: the proportion of children who 'seroconvert' to vaccine-serotypes after vaccination | 4-weeks post-primary series (approximately 18 weeks of age)
  The proportion of children with vaccine-serotype specific IgG antibody concentrations more than or equal to 0.35 mcg/ml after vaccination
The proportion of children with evidence of vaccine-serotype carriage | Approximately 18 months of age
  Vaccine-type carriage prevalence across arms
The proportion of children with evidence of vaccine-serotype carriage | Approximately 9 months of age
  Vaccine-type carriage prevalents across arms
The direct vaccine effectiveness of full/fractional doses of PCV13 against carriage of serotypes 6A and 19A | Approximately 18 months of age
  The direct effectiveness of full/fractional doses of PCV13 in preventing carriage of serotypes 6A and 19A compared to that of full dose PCV10
Opsonophagocytic activity of vaccine-induced antibody to 4 serotypes | Approximately 18 months of age
  Functionality of the antibody response

OTHER OUTCOMES:
Immunogenicity: the geometric mean concentration (GMC) of serotype-specific IgG | 4-weeks post-primary series (approximately 18 weeks of age)
  IgG GMCs elicited post-primary series
Safety: the prevalence of adverse events following immunisation by arm | Infants 6weeks-18 months of age
  The proportion fo children with adverse events following immunisation by arm
Immunogenicity: The geometric mean concentration (GMC) of serotype-specific IgG after the primary series of the 2p+1 schedule, prior to boost (9 months of age) and at the end of study follow-up at 18 months of age. | Approximately 9 and 18 months of age
  IgG GMCs at 9 and 18 months of age

CONTACTS AND LOCATIONS:
Overall Officials: J. Anthony G Scott, DTMH FMedSci, Principal Investigator — London School of Hygiene & Tropical Medicine, Keppel Street, London
Locations (1):
- KEMRI Wellcome Trust Research Programme, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The data will be open access and held in the LSHTM data repository (http://datacompass.lshtm.ac.uk/cgi/request_doc?docid=1); Data access will be granted upon reasonable request after the primary analyses of the trial, as specified, are published.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the primary analyses of the trial are published
Access Criteria: Upon reasonable request with pre-specified hypothesis
URL: http://datacompass.lshtm.ac.uk/cgi/request_doc?docid=1

REFERENCES:
- [Derived] Gallagher KE, Lucinde R, Bottomley C, Kaniu M, Suaad B, Mutahi M, Mwalekwa L, Ragab S, Twi-Yeboah L, Berkley JA, Hamaluba M, Karani A, Shangala J, Otiende M, Gardiner E, Mugo D, Smith PG, Tabu C, Were F, Goldblatt D, Scott JAG. Fractional Doses of Pneumococcal Conjugate Vaccine - A Noninferiority Trial. N Engl J Med. 2024 Nov 28;391(21):2003-2013. doi: 10.1056/NEJMoa2314620. Epub 2024 Sep 26. PMID 39330966

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03489018/Prot_SAP_ICF_000.pdf